CLINICAL TRIAL: NCT06685107
Title: Combination of Virtual Reality and Standard of Care Versus Standard of Care Alone for Acute Musculoskeletal Pain Management in Geriatric Emergency Department Patients: A Randomized Clinical Trial
Brief Title: Virtual Reality and Standard Care vs. Standard Care Alone for Acute MSK Pain in Geriatric ED Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-09-05
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Musculoskeletal Pain
Keywords: Geriatric; Emergency Medicine; Virtual Reality; Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Analgesia as determined by the treating physician
  Interventions: Other: Standard of Care Analgesia
- Virtual Reality (VR) + Standard of Care (SOC) (Active Comparator): Analgesia as determined by the treating physician and Virtual Reality experience that will use a geriatric-focused VR platform that has age appropriate VR content and will run for approximately 5-10 minutes
  Interventions: Other: Standard of Care Analgesia + Virtual Reality

INTERVENTIONS:
Other: Standard of Care Analgesia — Analgesia as determined by the treating physician
  Arms: Standard of Care (SOC)
Other: Standard of Care Analgesia + Virtual Reality — Analgesia as determined by the treating physician and Virtual Reality experience that will use a geriatric-focused VR platform that has age appropriate VR content and will run for approximately 5-10 minutes
  Arms: Virtual Reality (VR) + Standard of Care (SOC)

SUMMARY:
The proposed Virtual Reality as an Adjunct to Pain Management for Geriatric Patients in the ED (VRAP-ED) project will take place in the Emergency Medicine Department at Maimonides Medical Center. It seeks to enhance the analgesic practices for geriatric patients with acute painful conditions in the emergency setting. Although virtual reality (VR) has demonstrated effectiveness in reducing pain and anxiety in various clinical settings for juveniles and adults, the analgesic efficacy of VR for geriatric ED patients lacks established data. The project will use a geriatric-focused VR platform.

The project intends to improve pain management for almost 200 geriatric patients by evaluating the effectiveness of virtual reality (VR) in reducing pain and its impact on anxiety & stress reduction. The research project will conduct a randomized clinical trial to investigate the analgesic efficacy and impact on anxiety & stress by using VR as an adjunct to the standard of care (SOC) for pain management in elderly patients presenting to the ED with acute musculoskeletal pain. This will be investigated through a prospective, randomized, non-blinded clinical trial conducted over two years. Eligible patients will be randomly assigned to either the control (SOC) or intervention (SOC+VR) groups. The expected outcomes of this research study will provide insight into the feasibility of using VR in a busy emergency setting for one of the most commonly encountered painful syndromes and to assess the analgesic efficacy as well as the satisfaction of VR application by both patients and ED clinicians.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, randomized, non-blinded clinical trial, over a 2-year period, to investigate the efficacy of virtual reality (VR) on pain reduction as a primary outcome (quantitative outcome) and its effect on anxiety and stress (qualitative outcomes) as secondary outcomes in geriatric patients presenting to the ED of Maimonides Medical Center. This clinical trial will focus on patients with complaints of acute traumatic and non-traumatic musculoskeletal pain. These patients will be screened for eligibility and approached by study investigators. Upon meeting the eligibility criteria and completing an informed consent form, patients will be randomized into one of two study groups: 1) Standard of Care or 2) Standard of Care (SOC) plus Virtual Reality. Subjects will include geriatric patients, ages 65 and older, presenting to the ED with acute traumatic and non-traumatic musculoskeletal (MSK) painful syndromes with an initial numeric pain score of 4 and above on a standard 11 point (0 to 10) numeric rating scale (NRS) and requiring analgesia as determined by the treating ED physician. The total sample size for this trial will be 180 subjects (90 per group).

Eligible subjects in the trial will be randomized to either the control group or the intervention group. The control group will receive the standard of care (SOC) analgesia as determined by their treating physician and departmental guidelines. The intervention group will receive VR therapy via a headset as an adjunct to the SOC therapies prescribed. Study investigators will record pain scores, vital signs, and adverse effects at 0, 15, 30, 60, 90, and 120 minutes. In addition, anxiety and stress will be assessed before and after utilization of VR in the intervention group at 0, 30, 60 and 120 minutes. Subjects enrolled in the control group will have an evaluation of anxiety and stress recorded at 0, 30, 60, and 120 minutes as a part of secondary outcome measures as well.

ELIGIBILITY:
Inclusion Criteria:

* age of 65+
* Emergency Medicine patients
* non traumatic musculoskeletal painful condition
* pain score of 4+ on the numeric rating scale
* patient will warrant parenteral analgesia per treating physician
* patient will have to be awake, alert, and oriented to person, place, and time.
* comprehension of informed consent process and study related content
* ability to complete assessments

Exclusion Criteria:

* painful syndrome requiring emergent and/or urgent pain control
* altered mental status
* unstable vital signs
* history of recent epilepsy
* seizure disorder
* vertigo
* active headache
* nausea
* motion sickness
* dizziness

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 60 minutes
  A reduction of pain scores on the Numeric Rating Scale (0: no pain; 5 moderate pain; 10 extreme pain)

SECONDARY OUTCOMES:
Anxiety | 60 minutes
  Anxiety will be measured by the Spielberger State-Trait Anxiety Inventory (STAI-S) scale which range is between 20 and 80, with scores >40 indicative of appreciable anxiety.
Acute Stress | 60 minutes
  Acute Stress will be measured by 11-point stress Numerical Rating Scale (SNRS-11) (0 no stress; 5 moderate stress, 10: extreme stress) and at a self-reported nominal level
Adverse Effects | 60 minutes
  Adverse Effects occurring such as headache, dizziness, nausea, motion sickness

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT06685107/Prot_SAP_000.pdf